CLINICAL TRIAL: NCT04131816
Title: HeartHome: A Nurse-Driven, Home-Based Cardiac Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-2540
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome; ST-segment Elevation Myocardial Infarction (STEMI); Non-ST-Segment Elevation Myocardial Infarction (NSTEMI); Angina, Stable
Keywords: Cardiac Rehabilitation
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeartHome Intervention (Experimental): Participants will be in the HeartHome program for a total of 12 weeks.
  Interventions: Behavioral: HeartHome
- Control (No Intervention): De-identified data from 150 patients who attend a traditional cardiac rehabilitation program during the same general time of the HeartHome implementation

INTERVENTIONS:
Behavioral: HeartHome — The HeartHome program is an expanded home-based cardiac rehabilitation program that combines nurse home visits with telephone and electronic supports for participants that allows them to engage in cardiac rehabilitation activities at home.
  Arms: HeartHome Intervention

SUMMARY:
The purpose of this implementation trial is to execute a nurse-led, home-based cardiac rehabilitation (HBCR) program, evaluate the program's impact on patient outcomes over 6 months; and compare outcomes of HeartHome (HH) participants to a group of participants in traditional cardiac rehabilitation (CR).

DETAILED DESCRIPTION:
Despite being recognized as a class 1 recommendation by the American Heart Association (AHA), traditional CR is underused: only 20% of patients who need CR are referred, and only half of those referred enroll in the program. The primary barriers to enrollment in CR include the failure of providers to refer patients; systems that lack a clear, streamlined referral process; and patients who face multiple barriers, including knowledge, transportation, cost, time, and social-family support.

The HeartHome program is adapted from MULTIFIT, an evidence-based, interdisciplinary model of care developed at Stanford University was originally designed to provide coronary risk factor modification in post-MI patients, and later modified to implement consensus guidelines for providing HBCR to individuals with CVD using nurse managed care via telephone follow-up. HeartHome will combine nurse home visits with telephone and electronic supports for participants in a HBCR program that allows them to engage in cardiac rehabilitation programs at home.

In this trial, nurses will deliver the 12-week educational program to 150 participants. Participants will then complete follow-up assessments at the end of the program (3 months post enrollment), and then at 6-months post enrollment. The data collected will be compared to a control group that contains de-identified data from 150 patients that attend the traditional cardiac rehab program.

ELIGIBILITY:
Individuals are eligible for the HeartHome study if they meet all the following inclusion criteria:

* Diagnosed with one of the following conditions: myocardial infarction (MI)/acute coronary syndrome (ACS), ST-elevation myocardial infarction (STEMI), non-STEMI, percutaneous coronary intervention (PCI) or stable angina;
* Decline traditional cardiac rehab or do not respond to traditional cardiac rehab enrollment methods;
* Willing to have a nurse visit them in their home and receive follow-up phone calls and text messages for a 12-week intervention period;
* Understand the requirements of participation in and consent to the HeartHome program;
* Live within a 75-mile radius of the study site.

Individuals are not eligible for the HeartHome study if they meet any of the following exclusion criteria:

* Diagnosis of heart failure
* Diagnosis of valvular heart disease
* Presence of cardiac disease requiring surgery or other invasive procedure
* Impaired mental capacity resulting in an inability to understand or follow directions and study protocol
* Impaired functional abilities that prevent them from participating in physical activity
* Presence of any serious medical conditions that are likely to cause premature death or to impair functional capacity
* No access to a telephone

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Number of HeartHome patient referrals into the HeartHome program | 10 months after beginning of study
  Number of patient referrals into the HeartHome program will be measured by the total number of participants eligible to enroll in traditional cardiac rehab that were referred to the HeartHome program.
Proportion of HeartHome patient referral into the HeartHome program | 10 months after beginning of study
  Proportion of patient referrals into the HeartHome program will be measured by the number of patients referred to the HeartHome program relative to the number of patients referred to traditional cardiac rehab.
Proportion of HeartHome patient enrollments in the HeartHome program | 10 months after beginning of study
  Proportion of patient enrollments in the HeartHome program will be measured by the number of patients who enroll in the HeartHome program relative to the number of eligible patients referred to the HeartHome program. Enrollment is defined by signing the study consent form.
Participation in HeartHome's participants in-person visits | 12 weeks post HeartHome intervention start
  Participation in HeartHome's in-person visits will be measured by the number of in-person visits that each participant attends relative to the total number of in-person visits. The total number of visits possible per person is 5, with higher numbers associated with better participation.
Participation in HeartHome's participants interactive online classes | 12 weeks post HeartHome intervention start
  Participation in HeartHome's online classes will be measured by the number of online classes that each participant attends relative to the total number of interactive online classes. The total number of classes possible is 7, with higher numbers associated with better participation.
Participation in HeartHome intervention calls | 12 weeks post HeartHome intervention start
  Participation in HeartHome's calls will be measured by the number of calls that each participant attends relative to the total number of calls. The total number of calls possible is 8, with higher rate associated with better participation.
HeartHome intervention weekly goal adherence score | 12 weeks post HeartHome intervention start
  Adherence to weekly goals will be measured by participant goal achievement, which includes 33 opportunities for goal achievement and progression. The range is 0-33, with higher scores associated with greater adherence to weekly goals.
Number of sessions completed. | 13-weeks post start of HeartHome and control intervention
  Sessions completed by participants will be measured by the total number of calls, interactive online classes, and in-person visits attended. The total number of sessions is 20, with higher numbers associated with higher participation. Sessions completed by the control group will be measured by the total number of exercise sessions and classes attended. The total number of sessions for the control group is 46, with higher numbers associated with higher participation.

SECONDARY OUTCOMES:
HeartHome participants' physical function at baseline and at week 12 | 12 weeks post start of HeartHome intervention
  HeartHome participants' physical function will be measured by the six-minute walk distances at baseline and at 12 weeks. Longer distances (in meters) are associated with higher physical function.
Change in HeartHome participant's physical functioning, sub score of RAND SF-36 from baseline to week 12 and baseline to week 24. | 12- and 24-weeks post start of intervention
  Change in participants' physical function will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with better physical function.
Change in HeartHome participant's role limitations due to physical health, sub score of RAND SF-36 from baseline to week 12 and baseline to week 24. | 12- and 24- weeks post start of intervention
  Change in participants' role limitations due to physical health will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with fewer role limitations due to physical health.
Change in HeartHome participant's role limitations due to emotional problems, sub score of RAND SF-36 from baseline to week 12 and baseline to week 24. | 12- and 24- weeks post start of intervention
  Change in participants' role limitations due to emotional problems will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with fewer role limitations due to emotional problems.
Change in HeartHome participant's energy/fatigue, sub score of RAND SF-36 from baseline to week 12 and baseline to week 24. | 12- and 24- weeks post start of intervention
  Change in participants' energy/fatigue will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with higher energy/lower fatigue.
HeartHome participant's emotional well-being, sub score of RAND SF-36, assessed at baseline, week 12, and week 24. | 12- and 24-weeks post start of intervention
  Participants' emotional well-being will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with better emotional well-being.
HeartHome participant's social functioning, sub score of RAND SF-36, evaluated at baseline, week 12, and week 24. | 12- and 24-weeks post start of intervention
  Participants' social functioning will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with better social functioning.
HeartHome participant's bodily pain, a sub score of RAND SF-36, will be evaluated at baseline, week 12 and week 24. | 12- and 24- weeks post start of intervention
  Participants' bodily pain will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with less pain.
HeartHome participant's general health, sub score of RAND SF-36 at baseline, week 12, and week 24. | 12- and 24-weeks post start of intervention
  Participants' general health will be measured by a sub score of the RAND Short Form Survey Instrument (SF-36). The range is 0 - 100, and higher scores are associated with better general health.
HeartHome participant's change of participant and control physical functioning, sub score of RAND SF-36, from baseline to week 12 to end of program | 13-weeks post start of HeartHome and control intervention
  Participants' physical function will be measured by a sub score of the RAND SF-36. The range is 0-100, and higher scores are associated with better physical functioning.
HeartHome participant's blood pressure at baseline and weeks 3, 5, 7 and 12. | Baseline, weeks 3, 5, 7, and 12 of intervention
  Blood pressure will be measured by blood pressure measurements, measured in mmHg.
Participants' and control's blood pressure at baseline and 12 weeks | Baseline and 13-weeks post start of HeartHome and control intervention
  Blood pressure will be measured by blood pressure measurements, measured in mmHg.
Change in HeartHome participant's reported nicotine use from baseline to week 12 and baseline to week 24. | 12- and 24-weeks post start of intervention
  Rates of nicotine use will be measured by the change in participant-reported number of cigarettes smoked per week and patient-report of weekly frequency of non-cigarette nicotine use from baseline to week 12, and baseline to week 24.
HeartHome participant's waist circumference from baseline to week 12. | 12 weeks post start of intervention
  Waist circumference will be measured in centimeters at the beginning of the intervention (HeartHome program) and 12 weeks after beginning the intervention (HeartHome program). Negative changes in waist circumference are associated with greater weight loss.
HeartHome participant's Body Mass Index at baseline and week 12. | Baseline and 12 weeks post start of intervention
  Body Mass Index will be calculated from the participants' weights and heights at the beginning of the intervention (HeartHome program) and 12 weeks after beginning the intervention (HeartHome program). Lower numbers are associated with weight loss, and a patients' healthy range varies by age and gender.
Change of HeartHome participants' and control Body Mass Index from baseline to week 12 | Baseline and 13-weeks post start of HeartHome and control intervention
  Body Mass Index will be calculated by assessing participant weight and height at the beginning of the intervention (HeartHome program) and 12 weeks after beginning the intervention (HeartHome Program). Lower numbers are associated with weight loss, and a patients' healthy range varies by age and gender.
HeartHome participant's average weekly steps walked from baseline to week 12. | 12 weeks post start of intervention
  Average steps walked will be calculated using electronic fitness trackers at the beginning of the intervention (HeartHome program) and 12 weeks after beginning the intervention (HeartHome program). Higher numbers are associated with higher physical activity.
HeartHome participant's self-Reported and medical record reviewed number of hospital admissions 12 and 24 weeks after beginning of heart home program. | 12- and 24- weeks post start of intervention
  Participants' days of care utilization will be measured using the self-reported and medical record reviewed number of instances the participant is hospitalized in 12 and 24 weeks after the beginning of the heart home program.
HeartHome participant's self-Reported and medical record reviewed number of days hospitalized 12 and 24 weeks after beginning of heart home program. | 12- and 24- weeks post start of intervention
  Participants' days of care utilization will be measured using the self-reported and medical record reviewed number of combined days the participant spends in the hospital in 12 and 24 weeks after the beginning of the heart home program.
HeartHome participant and control number of hospital readmissions at 12 weeks | 13-weeks post start of HeartHome and control intervention
  Hospital readmission will be measured using patient self-reports and medical record reviews of hospital admissions (yes/no) at 12 weeks after the start of the intervention (HeartHome program).
HeartHome participant's self-reported and medical record reviewed number of ED visits without hospital admissions 12 and 24 weeks after beginning of HeartHome program | 12- and 24- weeks post start of intervention
  Participants' days of care utilization will be measured using the self-reported and medical record reviewed number of combined visits the participant makes to the Emergency Department (ED) in 12 and 24 weeks after the beginning of the heart home program.
HeartHome participant's self-reported and medical record reviewed number of specialist visits 12 and 24 weeks after beginning of the HeartHome program | 12- and 24- weeks post start of intervention
  Participants' number of specialist visits will be measured using self-reported and medical record reviewed number of combined cardiology visits 12 and 24 weeks after the beginning of the heart home program.
HeartHome participant's self-reported and medical record reviewed number of primary care visits 12 and 24 weeks after beginning of the HeartHome program | 12- and 24- weeks post start of intervention
  Participants' number of primary care visits will be measured using self-reported and medical record reviewed number of combined primary care visits 12 and 24 weeks after the beginning of the heart home program.
HeartHome participant's self-reported and medical record reviewed number of urgent care visits 12 and 24 weeks after beginning of the HeartHome program | 12- and 24- weeks post start of intervention
  Participants' number of urgent care visits will be measured using self-reported and medical record reviewed number of combined urgent care visits 12 and 24 weeks after the beginning of the heart home program.
HeartHome participant's Morisky 4-Item Scale scores at baseline, week 12, and week 24. | 12- and 24-weeks post start of intervention
  Management of participants' medications will be measured using the Morisky 4-item scale, which includes four questions to estimate the risk of medication non-adherence. The range is 0 to 4, and lower scores are associated with lower levels of medication adherence.
HeartHome participant's change in perceived stress scale from baseline to week 12 and baseline to week 24. | 12 and 24 weeks post start of intervention
  Participants' stress and emotional state will be measured using the perceived stress scale, which includes ten questions about individuals' feelings and thoughts during the last month. The range is 0-40, and higher scores are associated with higher levels of perceived stress.
HeartHome participant's change in dietary risk assessment from baseline to week 12 and baseline to week 24. | 12- and 24- weeks post start of intervention
  Participants' diet and lifestyle change will be measured by the dietary risk assessment, which includes 33 questions about how many servings of commonly eaten foods that participants eat in a usual day or an average week. The range is 0-52, higher scores represent a more healthful dietary pattern.
Participants' and control's dietary risk assessment scores from baseline to week 12 to dietary risk assessment scores of control group. | 13-weeks post start of HeartHome and control intervention
  Participants' diet and lifestyle change will be measured by the dietary risk assessment, which includes 33 questions about how many servings of commonly eaten foods that participants eat in a usual day or an average week. The range is 0-52, higher scores represent a more healthful dietary pattern.
HeartHome participant's change in PHQ-9 from baseline to week 12. | 12 weeks post start of intervention
  Participants' emotional state will be measured by the Patient Health Questionnaire (PHQ)-9, which includes 9 questions for screening, diagnosing, monitoring, and measuring the severity of depression. The range is 0 to 27, and scores represent cut-points for mild to severe levels of depression.
Change in participants' and control's PHQ-9 from baseline to week 12. | 13-weeks post start of HeartHome and control intervention
  Participants' emotional state will be measured by the PHQ-9, which includes 9 questions for screening, diagnosing, monitoring, and measuring the severity of depression. The range is 0 to 27, and scores represent cut-points for mild to severe levels of depression, with higher scores associated with more severe levels of depression.
HeartHome participant's change in New General Self-Efficacy score from baseline to week 12 and baseline to week 24. | 12- and 24-weeks post start of intervention
  Participants' confidence regarding task and situational performance is measured by the New General Self-Efficacy Scale, which includes 8 questions about participant confidence. The range is 8 to 40, and higher scores are associated with higher self-efficacy.
HeartHome participant's change in knowledge of cardiac rehabilitation from baseline to 12 weeks and baseline to 24 weeks. | 12- and 24-weeks post start of intervention
  Participants' knowledge of cardiac rehabilitation is measured by a 10-item Cardiac Rehabilitation Knowledge test at baseline, 12 weeks and 24 weeks. Scores range from 0-10, with higher scores associated with greater knowledge of cardiac rehabilitation.
Participants' and control's change in knowledge of cardiac rehabilitation from baseline to 12 weeks. | 13-weeks post start of HeartHome and control intervention
  Participants' knowledge of cardiac rehabilitation is measured by a 10-item Cardiac Rehabilitation Knowledge test at baseline, 12 weeks and 24 weeks. Scores range from 0-10, with higher scores associated with greater knowledge of cardiac rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Jones, PhD, RN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Health Care, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No